CLINICAL TRIAL: NCT00857259
Title: A Randomized, Double-masked, Parallel Group Study to Assess the Efficacy of Oral Everolimus, Either Alone or Added to Lucentis, in Patients With Neovascular Age-related Macular Degeneration
Brief Title: The Efficacy of Oral Everolimus in Patients With Neovascular Age-related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001A2203; EudraCT number: 2008-003550-15
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-07

CONDITIONS: Choroidal Neo-Vascular Age-onset Macular Degeneration; Age-related Macular Degeneration
Keywords: AMD; macular degeneration; Everolimus; Lucentis; Ranibizumab; Choroidal Neo-Vascular (CNV) age-onset macular degeneration; Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Everolimus; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Everolimus 5 mg (Experimental): 5 mg orally once daily plus sham ocular injection on Day 1 (Baseline) until Day 28
  Interventions: Drug: Everolimus
- Ranibizumab 0.5 mg (Active Comparator): Ranibizumab intra-vitreal therapy (IVT) 0.5 mg on Day 1 (baseline)
  Interventions: Drug: Ranibizumab
- Oral Everolimus (5mg) and Ranibizumab (0.5mg) (Active Comparator): Everolimus orally 5 mg once daily plus Ranibizumab Intra-vitreal therapy (IVT) 0.5 mg on day 1 (baseline)
  Interventions: Drug: Everolimus; Drug: Ranibizumab

INTERVENTIONS:
Drug: Everolimus — 5 mg oral tablet
  Arms: Everolimus 5 mg; Oral Everolimus (5mg) and Ranibizumab (0.5mg)
Drug: Ranibizumab — 0.5 mg administered by intravitreal injection
  Arms: Oral Everolimus (5mg) and Ranibizumab (0.5mg); Ranibizumab 0.5 mg

SUMMARY:
The study will assess the safety and efficacy of Everolimus (RAD001) alone or in combination with Lucentis in patients with neo-vascular age related macular degeneration (AMD)

ELIGIBILITY:
Inclusion Criteria:

* Patients with neovascular Age-Related Macular Degeneration (AMD)
* Best corrected visual acuity ( BCVA) of 20/40 or worse in study eye
* Patients with predominantly classic, minimally classic, or occult choroidal neovascularization in the macula of one eye (the study eye) who have had an inadequate response to VEGF inhibitors in the study eye. Inadequate response is defined as a gain of less than one line of visual acuity and persistent macular edema (central sub-fiel thickness ≥ 300 μm as measured by Optical Coherence Tomography (OCT) despite a minimum of 3 treatments with Lucentis or Avastin

Exclusion Criteria:

* Any concurrent ocular condition in the study eye that may result in substantial change in vision during the study
* Uncontrolled medical conditions such as cancer, angina, diabetes, viral or fungal infections, impaired lung function, history of stroke
* Patients who have macular edema in the study eye that, in the judgment of the investigator, is unlikely to respond to treatment. Examples of features that may guide the investigator's judgment about unresponsiveness are large regions of geographic atrophy, retinal angiomatous proliferation, or large regions of sub-retinal fibrosis. The presence of one of these features excludes a patient only if the investigator judges the study eye to have irreversible macular edema.
* active bacterial, fungal or viral infections at the time of enrollment, e.g. hepatitis B or C infection. Patients with risk factors for hepatitis B should be tested for hepatitis B viral load and serological markers at screening (a positive HBV-DNA, HBsAg). Patients with risk factors for hepatitis C should be tested using HCVRNA-PCR at screening. A clinical history of hepatitis B or hepatitis C will exclude the patient from the study.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (4):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Porter Adventist Hospital, Diagnostic Eye Laboratory, Denver, Colorado
  - Discover Vision Center, Independence, Missouri
- United Kingdom (8):
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Frimley
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford
  - Novartis Investigative site, Portsmouth
  - Novartis Investigative Site, Southampton
  - Novartis Investigator Site, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus 5 mg: 5 mg orally once daily plus sham ocular injection on Day 1 (Baseline)
- Everolimus and Ranibizumab: Everolimus oral 5 mg once daily plus ranibizumab Intra-vitreal therapy (IVT) 0.5 mg on day 1 (baseline)
Period: Overall Study
Arm/Group | Everolimus 5 mg | Ranibizumab 0.5 mg | Everolimus and Ranibizumab
Started | 8 | 1 | 7
Completed | 7 | 1 | 6
Not Completed | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus 5 mg | Ranibizumab 0.5 mg | Everolimus and Ranibizumab | Total
Number analyzed (Participants) | 8 | 1 | 7 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 75.9 (3.44) | 71.00 | 78.1 (14.23) | 76.6 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 6 | 9
  Male | 5 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Retinal Thickness From Baseline to Week 4, as Measured by Optical Coherence Tomography (OCT)
Description: Central retinal thickness was assessed by Optical coherence tomography (OCT). The primary thickness endpoint was the mean thickness of the foveal field of the macula map produced by the analysis of the sequence of six radial scans. Foveal field thickness was the average thickness of a circular field with a diameter of 1 mm. OCT images were analyzed by a central reading center.
Time Frame: Baseline and 4 weeks
Population: The Per Protocol Analysis Set (PPAS)consisted of all patients in the Full Analysis Set (FAS)who received study drug, completed the treatment phase of the trial without clinically significant protocol deviations and had non-missing central retinal thickness values for the study eye at both baseline and Day 28.
Measure: Mean (Standard Deviation); unit: µm
Groups:
- Oral Everolimus 5 mg: 5 mg once daily plus sham ocular injection on Day 1 (Baseline)
- Ranibizumab 0.5 mg: Ranibizumab intra-vitreal therapy 0.5 mg on Day 1 (baseline)
- Everolimus 5 mg and Ranibizumab 0.5 mg: Everolimus orally 5 mg once daily plus Ranibizumab intra-vitreal therapy (IVT) 0.5 mg on day 1 (baseline)
Arm/Group | Oral Everolimus 5 mg | Ranibizumab 0.5 mg | Everolimus 5 mg and Ranibizumab 0.5 mg
Number analyzed (Participants) | 6 | 1 | 6
µm
  Baseline | 454.8 (59.56) | 306.0 | 244.3 (80.37)
  Week 4 | 492.2 (122.16) | 308.0 | 217.6 (33.87)
  Change from Baseline | 37.3 (67.31) | 2.0 | -41.0 (56.18)

2. Secondary Outcome: Change in Visual Acuity From Baseline to Week 4 in Patients Treated With Everolimus
Description: Best corrected visual acuity (BCVA) was assessed on both eyes. BCVA measurements were taken in sitting position using Early Treatment Diabetic Retinopathy Study (ETDRs)-like visual acuity testing charts at an initial testing distance specific to test charts. BCVA is measured from the number of letters the patient can read on the eye chart.
Time Frame: Baseline and week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Groups:
- Everolimus 5 mg and Ranibizumab 0.5 mg: Everolimus oral 5 mg once daily plus ranibizumab Intra-vitreal therapy (IVT) 0.5 mg on day 1 (baseline)
Arm/Group | Everolimus 5 mg | Ranibizumab 0.5 mg | Everolimus 5 mg and Ranibizumab 0.5 mg
Number analyzed (Participants) | 6 | 1 | 5
Letters
  Baseline | 46 (16.91) | 67.0 | 55.3 (10.54)
  4 Weeks | 43 (17.09) | 69.0 | 63.2 (12.32)
  Change in baseline | -3 (7.59) | 2.0 | 4.4 (5.73)

ADVERSE EVENTS:
Description: Only two arms are represented in the Serious Adverse Events and Adverse Events > 5% Tables. The Ranibizumab 0.5 mg IVT arm is omitted because there were no SAEs or AEs reported in that treatment group.
Arm/Group | Oral Everolimus 5 mg | Everolimus 5 mg and Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 6/8 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Everolimus 5 mg (N=8) | Everolimus 5 mg and Ranibizumab 0.5 mg (N=7)
Lacrimation increased (Eye disorders) | 0 | 1
Macular degeneration (Eye disorders) | 1 | 0
Optic disc haemorrhage (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic wall hypertrophy (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or disclosure of the trial results in their entirety.